CLINICAL TRIAL: NCT00080158
Title: Treatment of Adolescent Suicide Attempters (TASA)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4623; U10MH066762 (NIH); U10MH066775 (NIH); U10MH066778 (NIH); U10MH066769 (NIH); U10MH066750 (NIH); DDTR B4-ARD; NCT00183534 (obsolete NCT alias)
Record Dates: First submitted 2004-03-24; First posted 2004-03-26 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Depression; Suicide, Attempted
Keywords: Dysthymic Disorder; Adolescent
MeSH Terms: conditions — Depression; Suicide, Attempted; Dysthymic Disorder | interventions — Fluoxetine; Sertraline; Citalopram; Escitalopram; Bupropion; Mirtazapine; Venlafaxine Hydrochloride; Lithium; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: fluoxetine
Drug: sertraline
Drug: citalopram
Drug: escitalopram
Drug: bupropion
Drug: mirtazapine
Drug: venlafaxine
Drug: lithium
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to compare the effects of three types of treatments for depressed teenagers who have attempted suicide.

DETAILED DESCRIPTION:
Suicide is the third leading cause of death in adolescents and is a major public health problem. Depression is the most common diagnosis for adolescent suicide attempts. Little is known about what treatment is best for these adolescents since they are usually excluded from participation in research studies.

Participants in this study will be randomly assigned to receive carefully monitored antidepressant medication with routine support and management, cognitive behavioral therapy (CBT), or a combination of antidepressant medication plus CBT.

ELIGIBILITY:
Inclusion Criteria:

* At least one suicide attempt or interrupted attempt within the past 45 days
* Continuously reside with a primary caretaker (parent, legal guardian, foster parent) for at least 6 months that can provide legal consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2004-03; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Greenhill, MD, Study Chair
Locations (6):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - New York University Child Study Center, New York, New York
  - Columbia University at the New York State Psychiatric Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Brent DA, Greenhill LL, Compton S, Emslie G, Wells K, Walkup JT, Vitiello B, Bukstein O, Stanley B, Posner K, Kennard BD, Cwik MF, Wagner A, Coffey B, March JS, Riddle M, Goldstein T, Curry J, Barnett S, Capasso L, Zelazny J, Hughes J, Shen S, Gugga SS, Turner JB. The Treatment of Adolescent Suicide Attempters study (TASA): predictors of suicidal events in an open treatment trial. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):987-996. doi: 10.1097/CHI.0b013e3181b5dbe4. PMID 19730274
- [Derived] Stanley B, Brown G, Brent DA, Wells K, Poling K, Curry J, Kennard BD, Wagner A, Cwik MF, Klomek AB, Goldstein T, Vitiello B, Barnett S, Daniel S, Hughes J. Cognitive-behavioral therapy for suicide prevention (CBT-SP): treatment model, feasibility, and acceptability. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):1005-1013. doi: 10.1097/CHI.0b013e3181b5dbfe. PMID 19730273